CLINICAL TRIAL: NCT05528575
Title: Randomised Three-arm Trial Investigating the Effects of Different Polyphenol and Prebiotic Combinations on Human Gut Microbiota and Perceived Cognitive State
Brief Title: Polyphenols, Prebiotics, the Gut Microbiome and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Glenn Gibson, Professor of Food Microbiology, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21/19
Record Dates: First submitted 2022-08-24; First posted 2022-09-06 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Stress, Psychological; Gut Bacteria
MeSH Terms: conditions — Stress, Psychological | interventions — blueberry extract; Tea; Chocolate; Inulin; Prebiotics; Polyphenols; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polyphenol (Experimental): Consume polyphenol combination for two weeks
  Interventions: Dietary Supplement: Blueberry, cranberry, green tea extract, cocoa
- Prebiotic (Experimental): Consume prebiotic combination for two weeks
  Interventions: Dietary Supplement: GOS, Inulin, RS2
- prebiotic and polyphenol (Experimental): Combination of prebiotics and polyphenols for two weeks
  Interventions: Dietary Supplement: prebiotics and polyphenols
- Placebo (Placebo Comparator): maltodextrin placebo for two weeks
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Blueberry, cranberry, green tea extract, cocoa — tablet supplements, available readily.
  Arms: Polyphenol
Dietary Supplement: GOS, Inulin, RS2 — Prebiotic combination, Inulin, GOS and RS2
  Arms: Prebiotic
Dietary Supplement: prebiotics and polyphenols — combination of the same prebiotics and polyphenols as above
  Arms: prebiotic and polyphenol
Dietary Supplement: Maltodextrin — maltodextrin, 10g per day
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate how different combinations of prebiotics and polyphenols affect the gut microbiota and perceived cognitive state. 40 volunteers will take part in this study who will be randomised into 4 different groups. One group will consume a placebo, whereas the other groups will consume prebiotics, polyphenols, or a combination of the two.

DETAILED DESCRIPTION:
* All participants will be asked to fill out a health screening questionnaire and inclusion/exclusion criteria will be reviewed for volunteer eligibility
* Valid informed consent will be obtained from the volunteer.
* Once the study begins, participants will be randomly allocated into 1 of 4 groups each assigned a different polyphenol or prebiotic product. the prebiotic content is dosed as follows: Inulin at 5g/d, GOS at 5g/d and Resistant Starch at 20g/d.
* Participants will be asked to consume their assigned product once per day. The length of the intervention is 14 days
* Participants will provide two stool samples: one on day 0 and one on day 14 of the study to identify changes in gut microbiota composition
* Urine samples will also be provided at day 0 and at day 14 looking for changes in urinary metabolites
* Participants will also be asked to fill out various mood related questionnaires on days 0 and 14 of the study.
* You will take your own blood pressure and heart rate on day 0 and day 14 and at least 3 times per week to try and link changes in gut microbiota composition with vascular health.
* Volunteers will be given containers and specimen pots to take home for initial and final faecal and urine collections. No treatment will be issued until initial stool and urine sample has been provided
* Maintenance of normal dietary patterns throughout the study is essential and participants will be required to complete food and drink logs throughout the study via a web-based app - on three consecutive days with one of the days being a weekend

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is healthy at the time of pre-examination
* Volunteer has high perceived stress levels (own self-assessment)
* Volunteer is aged ≥ 18 to ≤ 65 years at the time of pre-examination
* Volunteer is able and willing to comply with the study instructions
* Volunteer is suitable for participation in the study according to the investigator/study personnel
* Written informed consent is given by volunteer

Exclusion Criteria:

* No command of any local language
* Gastrointestinal disorders including IBS, IBD or other conditions that might affect the gut environment
* Food allergies or intolerances
* Using drugs (e.g. antibiotics) influencing gastrointestinal function (8 weeks before intervention)
* Use of laxatives
* Participants with any form of diagnosed diabetes (types I and II)
* Volunteers currently involved or will be involved in another clinical or food study
* History of drug (pharmaceutical or recreational) or alcohol abuse.
* participants are pregnant or are lactating
* Regular intake of probiotic or prebiotic supplements
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Bacteriology | baseline, pre-intervention, then After 14 days of intervention
  Changes in bacteriology
Mood Questionnaires | baseline, pre-intervention, then After 14 days of intervention
  various mood questionnaires

SECONDARY OUTCOMES:
Blood pressure | baseline, pre-intervention, then After 14 days of intervention. at least three times per week also
  Blood pressure taken systolic, diastolic and pulse

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom